CLINICAL TRIAL: NCT00568360
Title: Endoscopic Capillary Oximetry for Tumor Diagnosis in Head and Neck Cancer
Status: Terminated | Type: Observational
Why Stopped: Research cancelled; equipment broke
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: ENT0014; 79938 (Other: Stanford University Alternate IRB Approval Number); SU-11062007-817 (Other: Stanford University)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Oximeter

SUMMARY:
Endoscopy is a standard part of the evaluation of patients with head and neck cancer used for determining the extent of tumor involvement. However, not all areas involved by tumor are apparent visually. Preliminary results indicate that compared with normal tissues, tumors have abnormal levels of capillary oxygenation. The purpose of this study is to determine the ability of non-pulsatile visible light tissue oxygen monitoring to differentiate normal and tumor tissue based on capillary oxygenation during endoscopy Should this be possible, this method could be used to mark tumor extent and invasion, even when that invasion is up to 5mm blow the tissue surface.

ELIGIBILITY:
Inclusion Criteria:All patients with newly diagnosed head and neck cancer as well as those being seen for routine follow up with no evidence of current disease and healthy volunteers are eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with newly diagnosed head and neck cancer as well as those being seen for routine follow up with no evidence of current disease and healthy volunteers are eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2004-02; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Maxim PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States